CLINICAL TRIAL: NCT02513654
Title: An Open-label Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Repeat Dosing Lamotrigine in Healthy Chinese Subjects
Brief Title: Pharmacokinetics, Safety and Tolerability of Repeat Dosing Lamotrigine in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114536
Record Dates: First submitted 2015-07-30; First posted 2015-07-31 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Bipolar Disorder
Keywords: tolerability; repeat dosing; safety; healthy Chinese subjects; Pharmacokinetics; lamotrigine
MeSH Terms: conditions — Bipolar Disorder | interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lamotrigine dispersible tablets 25mg, 50mg, 100mg (Experimental): Each subjects will start dosing with lamotrigine 25mg dispersible tablet once daily at Day 1 and remain at this dose level for 2 weeks (Days1-14), then will be titrated to 50 mg once daily at Day 15 and last for weeks 3-4 (Days 15-28), and then titrated to 100 mg once daily at Day 29 during weeks 5-6 (Days 29-42).
  Interventions: Drug: Lamotrigine

INTERVENTIONS:
Drug: Lamotrigine — Lamotrigine dispersible tablets supplied in 3 different strengths 25 mg, 50 mg and 100 mg. These dispersible tablets appear as white or off-white tablets.

SUMMARY:
This Pharmacokinetic (PK) study is going to provide supplemental PK data for supporting bipolar Phase III study for New Drug Application (NDA) filing according to regulatory requirement. The primary objective of this study is to evaluate the PK of lamotrigine following repeat dosing of lamotrigine dispersible tablet in healthy Chinese subjects. This study consisted of Screening Phase (Days-14 to 0), Open-label Phase (Days 1 to 51) and follow-up Phase (10-17 days after last dosing). After signing the informed consent and confirm the eligibility, subjects will start dosing with lamotrigine 25 mg dispersible tablet once daily at Day 1 and remain at this dose level for two weeks (Days 1-14), then will be titrated to 50 mg once daily at Day 15 and last for weeks 3-4 (Days 15-28), and then titrated to 100 mg once daily at Day 29 during weeks 5-6 (Days 29-42). The total duration of the study will be approximately 10 weeks including screening and follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* Capable of returning to study site for follow-up according to requirement of protocol and willing to comply with the policy, procedure and restriction of the study. Capable of actively communicating with the investigator and completing the study-related documents; Capable of understanding the contents of the informed consent and signing a written informed consent prior to any study related procedures.
* Non-smoking Chinese healthy males or females as assessed by medical history and physical examination. Age 18-45 years (inclusive), at the time of signing the informed consent.
* Body weight >=50 kilogram (kg) and Body Mass Index (BMI) 19-24 kilogram per meter square (kg/m^2) (inclusive)
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator (in consultation with the GlaxoSmithKline (GSK) Medical Monitor if required) agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Aspartate transaminase (AST), Alanine transaminase (ALT), Alkaline phosphatase (ALP) and total bilirubin <= 1.5×upper limit of normal (ULN) (acceptable if only total bilirubin>1.5×ULN but direct bilirubin <35% of total bilirubin)
* No clinically significant abnormality on 12-lead electrocardiogram (ECG). Corrected QT interval (QTc) <450 millisecond (ms); or QTc <480 ms in subjects with Bundle Branch Block, based on single or averaged QTc values of triplicate ECGs obtained over a brief recording period.
* Normal blood pressure (systolic blood pressure 90-140 millimeter of mercury [mmHg], inclusive, diastolic blood pressure <90 mmHg) and heart rate (60-100 beats per minute [bpm], inclusive).
* A female subject with negative pregnancy test and not in lactating, and commit to take acceptable contraception measures during the study and in the 1 month post end of study.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy (for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records); or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 Milli-International Units per Mililiter (MIU/mL) and estradiol < 40 pico gram per milliliter (pg/mL) (<147 pico mole per liter [pmol/L]) is confirmatory]. Child-bearing potential with negative pregnancy test as determined by urine pregnancy test at screening or prior to dosing AND. Agrees to use one of the contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow-up visit. OR has only same-sex partners, when this is her preferred and usual lifestyle.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods after the first dose of study treatment and until the follow-up visit.

Exclusion Criteria:

* Unstable disease conditions; any laboratory measurements assessed by the investigator as clinically relevant (including ECG, hematology, biochemistry and urine analysis, etc.); Current or chronic history of cardiovascular, respiratory, gastrointestinal, endocrine, hematological, psychical or nervous system diseases, use of drug that can change the absorption, metabolism or elimination of study drug, or result in danger or other drugs or diseases that interfere with the interpretation of study data.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome and asymptomatic gallstones).
* Definite or suspected personal history or family history of adverse reactions or hypersensitivity to the study drug or to drugs with a similar chemical structure. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Subject with concurrent or previous neuropsychological disorders, as assessed by Columbia Suicidality Severity Rating Scale-Baseline Assessment or by the investigator, have suicidal tendency, or have committed suicidal behavior/attempt.
* Having any disease within 4 weeks prior to enrollment.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 14 days prior to the dosing day, which in the opinion of the Principal Investigator, may interfere with the study procedures or compromise safety.
* Drug or alcohol abuse or dependency within one year prior to enrollment. History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks. One drink is equivalent to 12 gram (g) of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Women of child bearing potential used oral or implanted contraceptives within the 30 days prior to study initiation, or received injections of chronically acting contraceptives in the 1 year prior to study initiation.
* Obvious evidence of active hematological diseases, or significant blood loss in the last 3 months.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of asthma, anaphylaxis or anaphylactic reactions, severe allergic responses.
* Subjects who have received lamotrigine previously (subjects who received placebo in a previous study will be allowed)
* Blood donation in the 3 months prior to enrollment. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* A positive Hepatitis B surface antigen (HBsAg) or positive Hepatitis C antibody (HCAb) result at screening
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) at screening.
* A positive test for syphilis at screening.
* Subject is mentally or legally incapacitated.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Other conditions which, in the Investigator's judgment, render patients unsuitable for the clinical study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-09-06 (Actual); Primary Completion 2015-11-11 (Actual); Study Completion 2015-11-11 (Actual)

PRIMARY OUTCOMES:
PK profile will be assessed by AUC (0-tau[24 hours]); Cmax; and accumulation ratios (Rcmax and Ro) following single and repeat dosing of lamotrigine dispersible tablet | Days 1, 14, 15, 28, 29, 42 and 44 to 51
  Blood samples for PK analysis will be collected on Days 1, 14, 28, and 42 before dosing (pre-dose) and at 0.5,1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 24 hours after administration. Other blood samples will be taken at 1 and 3 hours post dose on Day 15, and at 2 and 4 h post dose on Day 29. Additional blood samples will be taken at 48, 72, 96, 120, 168 and 216 hours after the administration of last dose on Day 42. Area under the concentration-time curve for a dose interval (AUC [0-tau{24 hours}]); observed maximum concentration (Cmax); and accumulation ratios (Rcmax and Ro) will be determined from the serum concentration-time data. Accumulation ratio will be calculated as follows: Ro = AUC(0-24) of Day14/AUC(0-24) of Day 1; and Rcmax = Cmax of Day14 / Cmax of Day 1

SECONDARY OUTCOMES:
PK profile will be assessed by Tmax; T1/2; Cssmax; Css,min; Css,avg; CL/F; and Vz/F and DF following single and repeat dosing of lamotrigine dispersible tablet. | Days 1, 14, 15, 28, 29, 42 and 44 to 51
  Blood samples for PK analysis will be collected on Days 1, 14, 28, and 42 before dosing (pre-dose) and at 0.5,1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 24 hours after administration. Other blood samples will be taken at 1 and 3 hours post dose on Day 15, and at 2 and 4 h post dose on Day 29. Additional blood samples will be taken at 48, 72, 96, 120, 168 and 216 hours after the administration of last dose on Day 42. Time to reach maximum concentration (Tmax), Terminal half-life (T1/2), Maximum concentration at steady state (Css,max), minimum concentration at steady state (Css,min), average steady state concentration (Css,avg), Apparent clearance (CL/F), Appearent volume of distribution (Vz/F), and Degree of fluctuation (DF) will be determined from the serum concentration-time data, as data permit.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Shanghai, China

REFERENCES:
- [Derived] Li Y, Zhang F, Xu Y, Hu J, Li H. Pharmacokinetics, Safety, and Tolerability of Lamotrigine Chewable/Dispersible Tablet Following Repeat-Dose Administration in Healthy Chinese Volunteers. Clin Pharmacol Drug Dev. 2018 Aug;7(6):627-633. doi: 10.1002/cpdd.449. Epub 2018 Mar 26. PMID 29578646
- See also: Results for study 114536 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/114536?search=study&b'search_terms=114536'#rs